CLINICAL TRIAL: NCT01369693
Title: In-vivo Extraction of Lead, Cadmium and Tobacco Specific Nitrosamines From Four Brands of Swedish 'Snus' in Regular Snus Users.
Brief Title: In-vivo Extraction of Pb, Cd and TSNA From Swedish Snus
Acronym: SMWS03
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Contract Research Organization el AB (Industry)
Collaborators: Swedish Match AB (Industry)
Responsible Party: Erik Lunell, MD, PhD, CROel AB
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2004/3
Record Dates: First submitted 2010-11-16; First posted 2011-06-09 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-06

CONDITIONS: Smoking Cessation; Smokeless Tobacco; Harm Reduction
Keywords: smokeless tobacco; Nicotine; Cadmium; lead; Tobacco Specific Nitrosamines
MeSH Terms: conditions — Smoking Cessation; Tobacco Use; Harm Reduction | interventions — Tobacco, Smokeless

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- General Portion 1 g pouch (Active Comparator)
  Interventions: Procedure: Buccal administration of nicotine
- Catch Licorice Portion 1 g pouch (Active Comparator)
  Interventions: Procedure: Buccal administration of nicotine
- Catch Licorice Portion Mini 0.5 g pouch (Active Comparator)
  Interventions: Procedure: Buccal administration of nicotine
- Catch Licorice Portion Dry Mini 0.3 g pouch (Active Comparator)
  Interventions: Procedure: Buccal administration of nicotine

INTERVENTIONS:
Procedure: Buccal administration of nicotine — Oral pouch, oral sachet, 0.3-1g, single dose. One pouch administered between upper lip and gum over 30 minutes
  Other Names: Smokeless Tobacco; ST; Potential reduced exposure products; PREP

SUMMARY:
In an open label, randomized, two-way cross-over study, 32 male healthy regular snus users will be given repeated doses of four different types of portion snus: "General", "Catch", "Catch Mini" and "Catch Dry Mini". Each portion of used snus will be collected and frozen (-20 oC) pending analysis of lead (Pb), cadmium (Cd), nicotine and tobacco specific nitrosamines (TSNAs). Unused snus is collected and deep frozen for analysis and calculation of extracted dose. Calculations of extracted amount of lead, cadmium, nicotine and tobacco specific nitrosamines (TSNAs) respectively, will be done for each type of snus.

DETAILED DESCRIPTION:
Comparisons:

A= "General Portion" 1 g portion snus containing approximately 8 mg nicotine per portion.

B= "Catch Licorice Portion" 1 g portion snus containing approximately 8 mg nicotine per portion.

C= "Catch Licorice Portion Mini" 0.5 g portion snus containing approximately 4 mg nicotine per portion.

D= "Catch Dry Licorice Portion Mini" 0.3 g portion snus containing approximately 4 mg nicotine per portion.

Swedish portion snus will be administered once every hour (4 administrations/brand) and will be kept between the upper lip and the gum for 30 minutes. Preload of own brand each morning.

ELIGIBILITY:
Inclusion Criteria:

* non-smokers, 18 to 50 years of age.
* Habitual use of > 7 portions snus daily since minimum 1 year.
* Healthy according to the health declaration and interview.
* Written informed consent given.

Exclusion Criteria:

* Concurrent participation in another clinical trial.
* History of allergy.
* History of allergy.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2004-05; Primary Completion 2004-08 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
In-vivo extraction of cadmium | 30 minutes' use
  Extracted amount = mean of 10 unused sachets - residual amount

SECONDARY OUTCOMES:
in-vivo extraction of tobacco specific nitrosamines (TSNAs)
  Extracted amount = mean of 10 unused sachets - residual amount in used sachet
In-vivo extraction of lead | 30 minutes' use
  Extracted amount = mean of 10 unused sachets - residual amount in one used sachet
In-vivo extraction of nicotine | 30 minutes' use
  Extracted amount = mean of 10 unused sachets - residual amount in one used sachet

CONTACTS AND LOCATIONS:
Overall Officials: Erik Lunell, MD, PhD, Principal Investigator — Croel AB
Locations (1):
- CROel AB, Helsingborg, Sweden